CLINICAL TRIAL: NCT07217379
Title: IGHID 12430 - Deliver-02 - A Phase 1, Open Label, Randomized Study To Evaluate The Safety And Tolerability Of MGD014 And MGD020 With A Latency Reversal Agent Versus Temporary Treatment Interruption In Persons With HIV-1 On Antiretroviral Therapy
Brief Title: The DART DELIVER-02 Study
Acronym: DELIVER-02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); US Military HIV Research Program (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-2690; HT94252430004 (Other Grant/Funding Number: Henry M Jackson Foundation, NIAID)
Record Dates: First submitted 2025-10-13; First posted 2025-10-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: HIV; latency reversal agent
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A - MGD014/MGD020 Infusions (Experimental): MGD014 and MGD020 infusions at Day 0, Week 2, Week 4 and Week 6.
  Interventions: Drug: MGD020; Drug: MGD014
- Arm B - MGD014/MGD020 Infusions with Temporary Treatment Interruption (TTI) (Experimental): MGD014 and MGD020 infusions at Day 0, Week 2, Week 4, and Week 6 in combination with a TTI from Day 4 to Week 8.
  Interventions: Drug: MGD020; Drug: MGD014; Other: Temporary treatment interruption
- Arm C - MGD014/MGD020 Infusions with Vorinostat (Experimental): MGD014 and MGD020 infusions at Day 0, Week 2, Week 8, and Week 10 in combination with VOR from Day 0 to Week 4 and Week 8 to Week 12.
  Interventions: Drug: MGD020; Drug: MGD014; Drug: Vorinostat

INTERVENTIONS:
Drug: MGD020 — Administered intravenously at 300mg/kg over 60 minutes.
Drug: MGD014 — Administered intravenously at 300mg/kg over 60 minutes.
Drug: Vorinostat — Administered orally at 400 mg every 72 hours.
  Arms: Arm C - MGD014/MGD020 Infusions with Vorinostat
Other: Temporary treatment interruption — Discontinuation of antiretroviral therapy (ART) through Week 8. If a participant meets protocol-defined ART restart criteria during the temporary treatment interruption (TTI), ART will be reinitiated immediately. Participants who do not meet restart criteria will remain off ART and continue weekly monitoring until Week 8, at which point ART will be resumed.
  Arms: Arm B - MGD014/MGD020 Infusions with Temporary Treatment Interruption (TTI)

SUMMARY:
This research study aims to find out how safe and well tolerated the experimental study drugs are when given to persons with HIV (PWH) taking antiretroviral therapy (ART). The study treatments are MGD014 and MGD020, which are two antibodies developed specifically for HIV, and Vorinostat, an oral medication to help expose HIV in cells to the antibodies. The study will measure the impact of study treatment on non-active HIV in cells, and how long MGD014 and MGD020 stay in the body after they are given.

In this study, participants will be randomly assigned to one of three groups. All participants receive MGD014 and MGD020, given sequentially as infusions through an IV for 4 doses. Participants in one group (group A) receive only MGD014 and MGD020. Participants in another group (group B) will stop taking their ART therapy for up to 8 weeks (a temporary treatment interruption (TTI)) while receiving MGD014 and MGD020. Participants in the third group (group C) receive Vorinostat in addition to MGD014 and MGD020. Total time of participation is about 8 months and involves 13 or 18 visits, depending on group assignment.

DETAILED DESCRIPTION:
This study is a phase 1, pilot, open-label study of MGD014 in combination with MGD020 in PWH on ART. The study is designed to characterize the safety, tolerability, pharmacokinetics (PK), and immunogenicity of the study drugs alone, and in combination with an latency reversal agent (LRA) or a TTI. Participants will be enrolled, undergo an initial evaluation and baseline sample collections, and then be randomized to 1 of 3 arms as follows:

Arm A: Continue baseline ART and receive biweekly MGD014/ MGD020 infusions at Day 0, weeks 2, 4 and 6.

Arm B: Initiate biweekly MGD014/ MGD020 infusions at Day 0 and undergo a TTI from Day 4 to week 8.

Arm C: Continue baseline ART, receive MGD014/ MGD020 infusions at Day 0, week 2, 8, and 10 in combination with VOR 400mg every 72 hours from Day 0 to week 4 and week 8-12

The study design will allow comparison of the impact of MGD014/MGD020 administration with continued ART alone, to MGD014/MGD020 administration with two different methods of latency reversal, 1) VOR, a latency reversal agent, and 2) TTI.

All participants will receive a total of 4 doses of MGD014/MGD020 at 300 mcg/kg administered as intravenous infusion. In Arms A and B, MGD014/MGD020 will be infused every 2-3 weeks. In Arm C, participants will receive two doses of MGD014/MGD020 at weeks 0 and 2, then again at weeks 8 and 10.In Arm C, participants will receive VOR 400 mg orally every 72 hours for 10 doses from Day 0 to week 4, and a second cycle of VOR 400 mg orally every 72 hours for 10 doses from week 8 to 12.

Study participants will have regular clinical assessments, including safety labs, viral load measurements, and CD4+ cell counts. Specimens will be stored for virologic and immunologic studies, including but not limited to comprehensive assessments of viral integrants, cell-associated HIV RNA, PK of MGD014/MGD020, and biomarkers of VOR exposure.

An independent safety monitor will provide study oversight and evaluate cumulative safety and other clinical data at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection initially documented by at least one of the following at any time prior to study entry:

   * any licensed rapid HIV test
   * HIV antibody test
   * HIV Ag/Ab assay

     …and documented confirmation by at least one of the following at any time prior to study entry:
   * licensed Western blot of HIV ½ antibody differentiation immunoassay
   * a second antibody test by a method other than the initial rapid HIV and/or HIV antibody assay
   * HIV-1 antigen, plasma HIV-1 RNA viral assay.
2. Ages ≥ 18 to ≤ 65 years old
3. Able and willing to give written informed consent.
4. Able and willing to stay in contact with site during the duration of the trial
5. Able and willing to provide adequate locator information.
6. Able and willing to comply with all study requirements through duration of the trial.
7. Continuous ART for a minimum of 24 months prior to screening, defined as not missing more than 9 consecutive days in the last 3 months prior to screening.
8. No change in any ART medication in the 30 days prior to screening.
9. Permitted ART regimens include:

   • At least 3 ART agents (not counting ritonavir or cobicistat as one of the agents if less than a 200 mg total daily dose). One of the agents must include an integrase inhibitor, NNRTI (Non-Nucleoside Reverse Transcriptase Inhibitors), or a boosted-PI (protease inhibitor).

   OR

   • Two (2) ART agents in which one of the agents is either a boosted protease inhibitor or an integrase inhibitor.

   Note: Other potent fully suppressive antiretroviral combinations will be considered on a case-by-case basis.
10. Participants must be determined to have an alternative ART regimen that can be constructed to assure availability of an effective option if assigned to Arm B and TTI leads to selection of virus resistant to the current regimen.
11. Ability and willingness of participant to continue ART throughout the study or temporarily discontinue ART for up to 8 weeks (for Arm B) under closely monitored supervision.
12. Plasma HIV-1 RNA <50 copies/mL at 2 time points in the 24 months prior to screening and never ≥50 copies/mL on 2 consecutive time points in the last 24 months.
13. No HIV RNA ≥200 copies/mL in the 6 months prior to screening.
14. CD4 cell count ≥ 400 cells/mm3 performed at screening.
15. At US sites, Hepatitis C (HCV) antibody negative result at screening or, if the participant is HCV antibody positive, a negative HCV RNA at screening; at Kenyan sites, participants must be HCV antibody negative at screening.
16. Hepatitis B surface antigen (HBsAg) negative at screening.
17. Women of child-bearing potential must have a negative serum pregnancy test with a sensitivity of at least 25 milli-international unit (mIU) per milliliter at screening Note: Women of child-bearing potential is defined as women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy
18. For participants with partners who do not have HIV or HIV status unknown, willingness to abstain from sexual intercourse, use a condom, and/or advise partner(s) to use pre-exposure prophylaxis (PrEP) consistently during the study TTI and until plasma HIV-1 RNA is <200 copies/mL if assigned to Arm B.
19. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) while on study and for 6 months after their last investigational product (IP) intervention.
20. All men and women participating in sexual activity that could lead to pregnancy must agree to consistently use at least one of the following forms of birth control for at least 21 days prior to Visit 3 (Day 0) and for 6 months after their last IP intervention.

    * Condoms (internal or external) with or without a spermicidal agent
    * Diaphragm or cervical cap with spermicide
    * Intrauterine device (IUD)
    * Tubal ligation
    * Hormone-based contraceptive
21. Agrees not to enroll on another study of an investigational agent during the study period, defined as any unlicensed investigational drug not yet approved for use in humans.
22. Willingness to defer live vaccinations (e.g., varicella, measles, mumps, rubella (MMR), yellow fever, oral polio, Mpox) from 30 days prior to enrollment through week 16.
23. Willingness to defer routine vaccination, including influenza, from 14 days prior to enrollment through Week 16 of the study.

    Note: Individuals who require vaccination will delay enrollment until 14 days after vaccination.
24. Agrees to refrain from blood donation during the course of the study.
25. Participants with Type 2 diabetes must have a hemoglobin A1C <8 or a fasting glucose ≤ 125 mg/dL; mmol/L at screening.
26. Adequate organ function as indicated by the laboratory values in Table 7 of the protocol.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Untreated syphilis infection defined as a positive rapid plasma reagin (RPR) without clear documentation of treatment.
3. Current treatment for HCV or HCV treatment within 6 months prior to enrollment.
4. Received any infusion blood product or hematopoetic growth factors within 3 months prior to enrollment.
5. Started ART within 90 days of diagnosis with acute HIV-1 infection.
6. Use of antiretrovirals that might interfere with MGD014 or MGD020: maraviroc (Selzentry), enfuvirtide (T-20), fostemsavir (Rubokia), Ibalizumab (Trogarzo).
7. Use of long-acting antiretroviral regimens given potential TTI.
8. Use of any of the following agents within 90 days prior to enrollment: immunomodulatory, cytokine, or growth stimulating factors such as systemic cytotoxic chemotherapy or immune globulin, interferons, coumadin, warfarin, or other Coumadin derivative anticoagulants.
9. Intent to use immunomodulatory treatment during the study.
10. Use of systemic corticosteroids within 30 days prior to enrollment, or anticipated need for periodic use of systemic corticosteroids during the study.

    Note: Participants receiving stable physiologic doses of glucocorticoids, defined as the equivalent of prednisone ≤10 mg/day, are not excluded.

    Participants receiving inhaled, intranasal, topical, intermittent intra-articular corticosteroids, or topical imiquimod are not excluded.

    Concomitant use of oral/systemic /intra-articular/inhaled/intranasal corticosteroids is prohibited for participants receiving ritonavir or cobicistat.
11. Use of the following medications that carry risk of torsade des pointes: amiodarone, arsenic trioxide, astemizole, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide, dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, probucol, procainamide, quinidine, sotalol, sparfloxacin, terfenadine, thioridazine.
12. Receipt of compounds with histone deacetylase (HDAC) inhibitor-like activity, such as valproic acid within the last 30 days. Potential participants may enroll after a 30-day washout period.
13. Use of any other investigational treatment within 6 months prior to enrollment, with the exception of Phase 2 or higher studies of antiretroviral agents.

    Note: Co-enrollment with other studies under an investigational new drug (IND) using an FDA approved medication that is not otherwise listed as prohibited will be considered on a case-by-case basis.
14. Any serious illness requiring systemic treatment or hospitalization, the participant must either complete therapy or be clinically stable on therapy, in the opinion of the site investigator, for at least 90 days prior to enrollment.
15. Any medical, psychiatric, substance abuse, occupational or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or assessment of safety.
16. History of malignancy within the last 3 years. Note: History of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary with documented resolution per topical treatment or complete resection determined by a dermatologist at least 3 months prior to enrollment.
17. Immune deficiency other than that caused by HIV infection.
18. Blood pressure consistently >150 mm Hg systolic and >100 mm Hg diastolic in the prior 6 months.
19. Grade 2 or higher QT prolongation as measured by corrected QT interval (QTc) as calculated by the Fridericia formula at screening.
20. History of acute or chronic pancreatitis.
21. Bleeding disorder including factor deficiency, coagulopathy or platelet disorder that requires special precautions (easy bruising without a formal diagnosis is not exclusionary) or chronic anticoagulation
22. History of pulmonary embolism or deep venous thrombosis.
23. History of hereditary angioedema, acquired angioedema or idiopathic angioedema.
24. Known allergy/sensitivity or hypersensitivity to components of study drugs.
25. Unstable asthma (e.g. sudden acute attacks occurring without an obvious trigger) or asthma requiring:

    1. Daily steroid or long-acting beta-agonist prevention
    2. Hospitalization in the last two years
26. Active chronic skin problems such as eczema or psoriasis not controlled with topical treatments.
27. Inability to communicate effectively with study personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants Experiencing At Least One Grade 3 or Greater Adverse Event that are Possibly or Definitely Related to Study Treatment | Day 0 through Week 8 (Arm A), Week 10 (Arm B), and Week 14 (Arm C)
  Safety data will include signs/symptoms, lab toxicities, and/or clinical events that are probably or definitely related to study treatment MGD014, MGD020, Temporary Treatment Interruption (TTI) and/or Vorinostat (VOR) through two weeks post completion of study treatment. The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 was used to measure safety where Grade 1 is defined as mild, Grade 2 is defined as moderate, Grade 3 is defined as severe, and Grade 4 is defined as potentially life-threatening.
Proportion of Participants who Received Full Course of Study Treatment | Day 0 through Week 6 (Arm A), Week 8 (Arm B), and Week 12 (Arm C)
  Receipt of the full course of study treatment is defined as receipt of all four MGD014 and MGD020 infusions. In addition for Arm B, the temporary treatment interruption (TTI) must have been longer than 10 days. In addition for Arm C, the participant must have received at least 16 Vorinostat (VOR) doses (Arm C).

SECONDARY OUTCOMES:
Serum PK Concentration of MGD020 | Day 0 through Week 26
  The concentration of MGD020 after infusions
Serum PK Concentration of MGD014 | Day 0 through Week 26
  The concentration of MGD014 after infusions
Incidence of Anti-drug Antibody (ADA) Formation to MGD020 | Day 0 through Week 24
  Number of participants who develop antibodies against MDG020
Incidence of Anti-drug Antibody (ADA) Formation to MGD014 | Day 0 through Week 24
  Number of participants who develop antibodies against MGD014
Number of Treatment Emergent Adverse Events (TEAEs) | Day 0 through Week 26
  Safety data will include signs/symptoms, lab toxicities, and/or clinical events.
Number of Serious AEs (SAEs) | Day 0 through Week 26
  Safety data will include signs/symptoms, lab toxicities, and/or clinical events.
Number of Adverse Events Leading to Treatment Discontinuation | Day 0 through Week 26
  Safety data will include signs/symptoms, lab toxicities, and/or clinical events.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L. Gay, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- University of North Carolina, Chapel Hill, North Carolina, United States
- Kenya (2):
  - Moi University Clinical Research Center, Eldoret
  - Kenya Medical Research Institute/Walter Reed Project, Kericho

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months after publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.
URL: http://www.unc.edu